CLINICAL TRIAL: NCT06747650
Title: Dialectical Behavior Therapy for Adolescents With Fetal Alcohol Spectrum Disorders Feasibility Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Christie Petrenko, Research Associate Professor, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00009819; 1F31AA031596-01 (NIH)
Record Dates: First submitted 2024-12-18; First posted 2024-12-24 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Fetal Alcohol Spectrum Disorder
MeSH Terms: conditions — Fetal Alcohol Spectrum Disorders | interventions — Dialectical Behavior Therapy

STUDY DESIGN:
Intervention Model Description: A single cohort of teens with FASD will be administered DBT-A for the purpose of feasibility testing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active DBT-A Intervention Arm (Experimental): A single cohort of teens with FASD will be administered DBT-A for the purpose of feasibility testing.
  Interventions: Behavioral: Dialectical Behavior Therapy for Adolescents

INTERVENTIONS:
Behavioral: Dialectical Behavior Therapy for Adolescents — Standard of care (SOC) DBT-A includes approximately six weeks of pretreatment, and approximately six months of DBT-A skills group, individual therapy, and 24/7 phone coaching. During pre-treatment, clients are oriented to the DBT-A model and client commitment to treatment is established. After approximately six weeks, the client enters DBT-A skills group along with their caregiver. This skills group meets weekly for 1.5 hours and clinicians explain the five main DBT-A skills (mindfulness, distress tolerance, emotion regulation, interpersonal effectiveness, and walking the middle path) via PowerPoints and discussion. Clients and their caregivers are assigned weekly homework. At the same time, teens are completing weekly 1-hour individual therapy sessions where they are utilizing the skills learned in group. Both teens and caregivers have access to what DBT-A calls 24/7 phone coaching. This phone coaching is 24/7 access to a therapist when a crisis is arising.

SUMMARY:
The purpose of this study is to test the feasibility of dialectical behavior therapy for adolescents (DBT-A) with fetal alcohol spectrum disorders (FASD). In partnership with a community mental health practice, Genesee Valley Psychology (GVP), two cohorts of five adolescents with FASD and their caregivers will participate in an already existing comprehensive DBT-A program (including individual therapy, group skills training, and 24/7 phone coaching). This program has been adapted for neurodivergent teens, including the development of trainings for mental health clinicians on FASD. The aim of the current study is to assess the acceptability of DBT-A from the perspective of teens, caregivers, and clinicians. Additionally, barriers and facilitators of implementing DBT-A with teens with FASD, as well as the feasibility of the research protocol will be assessed to inform later larger-scale trials.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:

For adolescents:

* Ages 14-17 years
* Have a diagnosis of FASD under any diagnostic criteria
* Residing in the state of New York
* Willing and able to attend group sessions virtually
* Have one of the following:

  1. A diagnosis of disruptive mood dysregulation disorder, borderline personality disorder, or multiple other serious mental health diagnoses
  2. A history of multiple psychiatric hospitalizations and/or recurring presentation at psychiatric emergency rooms
  3. A score of 7+ on the McLean screening instrument (MSI; instrument attached and included in eligibility screen)
* Have functional deficits in three of five problem areas:

  1. Emotional dysregulation
  2. Impulsivity (including avoidance)
  3. Interpersonal challenges
  4. Teenager and family challenges
  5. Reduced awareness and focus
* Access to the internet and device with Zoom capabilities

For caregivers:

* Parent or legal guardian of an adolescent (ages 14-17 years) with an FASD diagnosis
* Residing in the state of New York
* Willing and able to attend group sessions virtually
* Access to the internet and device with Zoom capabilities

For clinicians:

* Employee of GVP
* Administered DBT-A to teens with FASD as part of this study

Exclusion Criteria:

* • Adolescent, caregiver, or clinician has insufficient proficiency in English

  * Primary psychotic disorder
  * Ongoing substance/drug dependence or eating disorder at such a level that would impede engagement with DBT modalities (i.e. if an individual requires detoxification or hospitalization for stabilization)
  * Adolescent or caregiver has a moderate to severe intellectual disability (IQ < 51)

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2024-12-24 (Actual); Primary Completion 2025-10-29 (Actual); Study Completion 2025-10-29 (Actual)

PRIMARY OUTCOMES:
Difficulties in emotion regulation scale caregiver and self-report | Baseline and Week 35
  The Difficulties in Emotion Regulation Scale (DERS) is a validated self-report measure designed to assess challenges in regulating emotions. It evaluates six dimensions of emotion regulation difficulties: non-acceptance of emotional responses, difficulties engaging in goal-directed behavior when distressed, impulse control challenges during emotional distress, lack of emotional awareness, limited access to effective emotion regulation strategies, and lack of clarity about emotional experiences. This study will utilize the brief form consisting of 18 items rated on a Likert scale, with higher scores indicating greater difficulties in emotion regulation. Each scale has a score range of 3 to 15.
Child behavior checklist caregiver and youth report | Baseline and week 35
  The Child Behavior Checklist (CBCL) is a standardized, parent-reported questionnaire designed to assess a wide range of emotional and behavioral problems in children and adolescents. It is part of the Achenbach System of Empirically Based Assessment (ASEBA) and evaluates competencies and problems in various domains. The CBCL yields scores across internalizing behaviors (e.g., anxiety, depression), externalizing behaviors (e.g., aggression, rule-breaking), and total problems. It also provides syndrome scales (e.g., anxious/depressed, somatic complaints, social problems) and DSM-oriented scales aligned with diagnostic criteria. The scales are reported as t-scores with a mean of 50 and a standard deviation of 10. The higher the t-score, the more significant the behavioral issues.
The theoretical framework of acceptability questionnaire | Week 35
  The Theoretical Framework of Acceptability (TFA) defines acceptability as a multi-dimensional construct. The TFA identifies several dimensions that shape individuals' experiences with an intervention, including their affective attitude toward the intervention, the perceived burden or effort required to engage with it, the alignment of the intervention with their personal values and beliefs, and the extent to which they understand its purpose and mechanisms. It also considers the perceived opportunity costs of participation, participants' beliefs about the intervention's effectiveness, and their confidence in their ability to successfully engage with it. Each question is a 5-point Likert scale, with higher scores indicating highter acceptability of treatment.

SECONDARY OUTCOMES:
Patient Health Questionnaire 9-item | Base line to 9 months
  The Patient Health Questionnaire-9 (PHQ-9) is a widely used self-report tool designed to screen for, diagnose, and monitor the severity of depressive symptoms. It is based on the diagnostic criteria for major depressive disorder outlined in the DSM, making it a clinically relevant and psychometrically robust measure. The PHQ-9 consists of nine items that assess the frequency of core depressive symptoms, such as low mood, loss of interest or pleasure in activities, fatigue, changes in sleep or appetite, feelings of worthlessness, difficulty concentrating, and thoughts of self-harm or death. Respondents rate the severity of these symptoms over the past two weeks on a four-point scale, ranging from "not at all" to "nearly every day," yielding a total score that indicates depression severity. Higher scores suggest more severe depressive symptoms.
General Anxiety Disorder 7-item | Base line to 9 months
  The Generalized Anxiety Disorder 7-item scale (GAD-7) is a brief, self-report measure designed to screen for, assess, and monitor the severity of generalized anxiety symptoms. It evaluates core symptoms of anxiety based on criteria outlined in the DSM, including excessive worry, restlessness, difficulty concentrating, irritability, muscle tension, and sleep disturbance. Respondents rate the frequency of these symptoms over the past two weeks on a four-point Likert scale, ranging from "not at all" to "nearly every day." The total score provides an indication of anxiety severity, with higher scores reflecting greater symptom burden.
Clinician therapeutic note documentation | Base line to 9 months
  Clinician documentation of client participation, homework completion, attention during session, camera use during virtual sessions, and therapy-interfering behaviors.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No